CLINICAL TRIAL: NCT00181181
Title: The Effect of Statin Use on Vascular Function in Hypertensive Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Coronary flow by echo Doppler was obtainable in about 50% of subjects. The study was stopped early because of insufficient sample size to achieve adequate power
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other); Procris Pharmaceuticals (Industry)
Responsible Party: Pamela Ouyang MBBS, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HBV03-03-03-02
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2006-09

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Atorvastatin (Active Comparator): Atorvastatin for 3 months
  Interventions: Drug: atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: atorvastatin — Atorvastatin 80 mg daily for 3 months
  Arms: Atorvastatin
Other: placebo — placebo daily
  Arms: Placebo

SUMMARY:
This research is being done to find if treatment with atorvastatin, a drug that reduces cholesterol, improves the function of blood vessels among people with high blood pressure. Adults with mildly high blood pressure, or who are taking medication for high blood pressure but are otherwise healthy may join, with the approval of their health care provider. The study period is 14-17 weeks. Approximately 50 to 60 subjects will take part in the study.

DETAILED DESCRIPTION:
Subjects will be treated with either atorvastatin or placebo. We will test the function of the blood vessels at baseline and after 3 months of treatment. Treatment of people with high blood pressure with atorvastatin is experimental. It is necessary to compare the experimental treatment with placebo to know if it works. Subjects will be assigned to a group given the experimental treatment or placebo by chance (like flipping a coin). Subjects will be evaluated for heart, lung, kidney or liver disease. Only people without any of these diseases may join the study.

Screening visit:

Subjects will be asked to fast overnight before the screening visit. Chest Examination and EKG: On the first visit, we will perform a chest examination and an EKG. The subject's blood pressure will be measured several times, with 2 minutes between measurements after the subject has sat quietly for several minutes.

Exercise Stress test: Subjects will be scheduled to have an exercise treadmill test which consists of walking on a moving platform. Your heart rate, blood pressure and EKG will be watched while you exercise. The speed and slope of the platform will be increased to cause a gradual increase in the workload. The EKG during exercise will show if there is good blood supply to the heart.

Urine test for pregnancy: This test will be done for women of childbearing age who are of child bearing potential.

Blood tests: We will draw 15 ml (about 1 tablespoonful) of blood for tests of cholesterol, glucose, liver and kidney function. After tests are completed during the screening visit, subjects are given advice about diet and healthy lifestyle to control blood pressure. The screening results will indicate whether a subject should not join this study. If there are any abnormal results, the investigators will refer the subject to their primary health care provider. The total amount of time required for the screening visit is two hours.

If subjects qualify for joining the study, a baseline visit will be scheduled within 2 weeks. If a subject meets all conditions, except that the blood pressure is too high or if they are taking a blood pressure medication not allowed by the study, their health care provider will be contact for permission to give a blood pressure medication that is allowed. If the subject is given blood pressure medication, a follow-up visit after two weeks will be scheduled to check the blood pressure.

Blood pressure check visit:

This visit is scheduled only if blood pressure medication has been added or changed. The blood pressure will be measured several times, with 2 minutes between measurements. If the blood pressure is controlled, the subject may continue in the study. The baseline visit will be scheduled within 2 weeks.

Baseline visit: Subjects will be asked to not take any medication for 24 to 48 hours before the visit and may not eat any food, or drink any coffee, tea, milk, citrus fruit juice or caffeinated soda for 8 hours before the tests. Pulse Pressure will be recorded after sitting quietly at rest. The blood pressure will be measured several times, with 2 minutes between measurements.

Urine tests: Urine will be collected to test its chemistry. Brachial artery reactivity: The subject will lie on a bed. The blood pressure is measured in one arm.Another blood pressure cuff will be wrapped around the other arm. The artery of the arm will be studied using an echo machine that uses sound waves to image the blood vessel. The blunt tip of the echo probe will be placed on the arm after applying gel to the skin. Images of the artery will be recorded for two minutes. The cuff is then inflated and will squeeze the arm tightly for five minutes and will then be released. Images of the artery will be made throughout the five minutes while the cuff is inflated and for three minutes after the release of pressure. During the test the pulse in the fingers of the hands will be recorded using two finger straps.

Pulse Wave Velocity: The investigators will use an echo machine to measure how fast the pulse travels between the subject's neck and thigh. For this test the subject will lie down and a technician will hold one echo probe on the neck and one on the upper thigh.

Blood tests: At this visit 15 ml (about 1 tablespoonful) of blood will be drawn for tests of insulin, markers of inflammation and platelet function.

Coronary Artery Flow Velocity Reserve: The subject will lie on a bed and a fine tube (an i.v. line) will be placed in the arm to allow study drugs to be injected into the vein. A drug that will make blood vessels clearly visible by echo will be injected in your vein. An echo technician will place the tip of the echo probe on the chest after applying gel to it. The technician will record images of your heart for 10 minutes. Then adenosine, which increases the blood flow to the heart, will be injected into the vein, and echo images will be recorded for the next 5 minutes. Adenosine is a drug that is used clinically in stress tests. Subjects may feel a desire to take deep breaths as if they had performed strenuous exercise. In all, the drug that will make the arteries clearly visible will be injected 10 minutes before adenosine and 5 minutes with adenosine for a total of 15 minutes. The i.v. drugs will be stopped after the recording. EKG will be monitored throughout the procedure. Subjects may request that the i.v. drugs and the recording be stopped they are very uncomfortable. The blood flow reserve can be measured later from these recorded images.

The total time spent for the tests during the baseline visit is two hours and thirty minutes.

Skin Cholesterol Measurement: Prior to the skin test the hands are washed. The palm of the hand will also be cleaned with an alcohol pad. A small amount of cholesterol binding solution will then be placed on the palm of the hand for 1 minute. This will then be blotted off. An indicator solution will then be placed in the same area for 2 minutes. This will result in the development of a spot of blue color. The blue color can be wiped off with a paper towel at the end of the test. A handheld spectrophotometer (a small device that can "read" the color intensity on the skin where the solution was placed) will be placed against the palm. This device is attached to a laptop computer that will generate a numerical skin cholesterol value. A sample of the cells from the skin surface will be collected by pressing a piece of sticky tape 10 times on each of the subject's palms. The tape is about as sticky as that used for office stationery. This tape will be sent to another laboratory for analysis.

Dispensing of drug: Subjects will then be given a packet of medication to be taken over the next three months. Subjects will take one capsule each day.

Final Visit: The final visit will be scheduled 3 months following the baseline visit. Subjects may not take any medication for 24 hours before the visit and may not eat any food, or drink any coffee, tea, milk or caffeinated soda for 8 hours before the visit. All the tests performed at the baseline visit will be repeated. Approximately 30 ml (about 2 tablespoonsful) of blood will be drawn for tests including cholesterol, glucose, insulin, liver and kidney function, and markers of inflammation. Urine will be collected for urine tests. The total time spent for the tests during the final visit is two hours and thirty minutes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 20-75 years of age.
* The subjects will have a sitting systolic blood pressure measurement of 140-159 mm Hg (measured using JNC VI procedures) OR a prescription verified history of the use of stable (for 3 months) antihypertensive medication (certain drugs are excluded below). Potential subjects not on therapy who have a systolic BP of 140-159 mmHg will be advised on diet and lifestyle changes according to JNC VI guidelines prior to study participation.
* They must be able to give informed consent.

Exclusion Criteria:

* Subjects currently using lipid-lowering medication such as statins, niacin or gemfibrozil.
* Systolic BP > 159 mmHg or diastolic BP > 99 mmHg despite anti-hypertensive medication. Subjects who have blood pressure readings above these values will be given a trial of antihypertensive therapy for two weeks using the drugs hydrochlorthiazide and/or metoprolol with permission from them and their primary healthcare provider. If controlled, they will be allowed to enroll.
* Subjects on clonidine. Subjects on clonidine who express interest in the study will be considered if their primary health care provider permits the investigators to change them on to allowed antihypertensive medication, i.e., hydrochlorthiazide or metoprolol, and they meet enrollment criteria after two weeks of therapy.
* Subjects on ACE inhibitors or calcium channel blockers who express interest in the study will be considered if their primary health care provider permits the investigators to change them on to allowed antihypertensive medication, i.e., hydrochlorthiazide or metoprolol, and they meet enrollment criteria after two weeks of therapy. If beta-blocker/diuretic treatment is not effective or not tolerated, or if advised by the subject's primary health care provider, subjects may remain in the study on ACE inhibitors or calcium channel blockers.
* Subjects being treated with antifungal agents or the antibiotic erythromycin.
* Women using oral contraceptive drugs.
* Diabetic patients that are not on antihypertensive medication.
* Subjects who have EKG abnormalities during the screening visit, ischemic EKG abnormalities on stress testing, or history of prior diagnosis of ischemic heart disease, or use of digoxin, nitroglycerine/anti-anginal agents, theophylline-like drugs or antiarrhythmic medication.
* Subjects with a history of chronic obstructive airway disease, or evidence of such disease at clinical examination during the screening visit. (x) Persons who are current smokers.
* Subjects with abnormal liver and renal function tests at screening visit. - Women who are pregnant (by history or pregnancy test) or are planning pregnancy during the study period, or are nursing infants.
* Persons with severe obesity defined as BMI > 40 kg/m2.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-05; Primary Completion 2006-06 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of statin therapy on vascular function,on coronary microvascular function, on markers of inflammation and NO metabolites ,and on skin cholesterol of hypertensive subjects. | 3 months
  microvascular function by echo doppler of coronary flow

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Ouyang, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States